CLINICAL TRIAL: NCT01120834
Title: Phase I/II Study of 5-azacitidine in Combination With Vorinostat in Patients With Relapsed or Refractory DLBCL
Brief Title: Study of 5-azacitidine in Combination With Vorinostat in Patients With Relapsed or Refractory Diffuse Large b Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0912010795
Record Dates: First submitted 2010-04-19; First posted 2010-05-11 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: diffuse large b cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Azacitidine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental)
  Interventions: Drug: azacytidine; Drug: vorinostat

INTERVENTIONS:
Drug: azacytidine — * Dose level 1: azacitidine 55 mg/m2 on days 1-5
  * Dose level 2: azacitidine 75 mg/m2 on days 1-5
  * Dose level 3: azacitidine 55 mg/m2 on days 1-5
  * Dose level 4: azacitidine 75 mg/m2 on days 1-5
  Each cycle = 28 days. Subjects may receive up to 6 cycles.
Drug: vorinostat — * Dose level 1: oral vorinostat at 300 mg BID on Days 1-7.
  * Dose level 2: oral vorinostat at 200 mg BID on Days 1-7.
  * Dose level 3: oral vorinostat at 300 mg BID on Days 1-14.
  * Dose level 4: oral vorinostat at 200 mg BID on Days 1-14.
  Each cycle = 28 days. Subjects receive up to 6 cycles.

SUMMARY:
This will be a phase I/II study of 5-azacitidine in combination with vorinostat in patients with relapsed or refractory DLBCL. Combination therapy with methyltransferase inhibitors and histone deacetylase inhibitors is highly synergistic in DLBCL cells, and both classes of drugs can also synergize powerfully with standard anti-lymphoma chemotheraputics such as doxorubicin in pre-clinical studies. We hypothesize that azacytidine + vorinostat combination therapy will be safe and effective in selected patients with relapsed or refractory DLBCL. We also hypothesize that patients demonstrating objective responses to this combination therapy display specific epigenetic signatures, and that a biomarker or gene classifier can be generated which will identify those patients likely to respond.

DETAILED DESCRIPTION:
Eligible subjects will have biopsy proven relapsed or refractory DLBCL, have preserved hematologic and other organ function, and have either progressed following or be inappropriate candidates for autologous stem cell transplantation.

Patients will be treated with 5-azacitidine via subcutaneous administration and vorinostat orally at four different dose levels as described below:

* Dose level 1: azacitidine 55 mg/m2 on days 1-5 and oral vorinostat at 300 mg BID on Days 1-7.
* Dose level 2: azacitidine 75 mg/m2 on days 1-5 and oral vorinostat at 200 mg BID on Days 1-7.
* Dose level 3: azacitidine 55 mg/m2 on days 1-5 and oral vorinostat at 300 mg BID on Days 1-14.
* Dose level 4: azacitidine 75 mg/m2 on days 1-5 and oral vorinostat at 200 mg BID on Days 1-14.

Each cycle will be of 28 days and patients will be treated for up to 6 cycles.

Up to 8 patients will be enrolled at each dose level. If at any time 2 patients in a given cohort experience DLT, enrollment to that level will be discontinued.

Efficacy will be assessed by standard radiographic and other criteria at baseline and at the end of treatment to determine ORR. Patients will be followed for 2 years or until disease progression.

Tumor samples will be obtained for correlative studies at baseline through core needle or surgical biopsy, with an additional biopsy performed on day 15 of cycle 1 as a pharmacodynamic endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diffuse large B cell lymphoma, relapsed after or resistant to prior systemic therapy.
* Subjects must have measurable disease on cross sectional imaging that is at least 1.5 cm in diameter.
* Patients should have relapsed following or be deemed ineligible for autologous stem cell transplantation. There is no limit to number of prior therapies.
* Age > = 18 years.
* ECOG performance status < = 2.
* Patients must have normal organ and marrow function as defined below:

  * ANC > = 1,000/uL
  * platelets > = 75,000//uL
  * total bilirubin < = 2 X upper limit of normal
  * AST(SGOT)/ALT(SGPT) < = 2.5 X upper limit of normal
  * Serum creatinine < = 1.5 X upper limit of normal (ULN)
* Women of childbearing potential must have a negative serum pregnancy test prior to treatment
* The effects of these investigational agents on the developing human fetus at the recommended therapeutic doses are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A woman who becomes pregnant while participating in the study must withdraw from the study immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior allogeneic transplant
* Patients may not be receiving any other investigational agents.
* Patients may not have previously received anti-lymphoma therapy with an HDAC inhibitor (.e.g. Depsipeptide, MS-275, LAQ-824, PXD-101, and valproic acid). Patients who have received an HDAC inhibitor for another indication such as epilepsy may enroll after a 30-day washout period
* Patients with known active CNS lymphoma. Subjects with previous CNS lymphoma that have been treated with chemotherapy, radiotherapy or surgery who have remained asymptomatic for 90 days (3 months) and demonstrate, no CNS lymphoma, as shown by lumbar puncture, CT scan or MRI, are eligible..
* Patients with known hypersensitivity to azacytidine, vorinostat or mannitol.
* Patients with a currently active second malignancy.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* QTc interval > 0.470. Consider discontinuation of medications that prolong QTc interval to eliminate this exclusion if medically appropriate.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: azacytidine: • Dose level 1: azacitidine 55 mg/m2 on days 1-5
  * Dose level 2: azacitidine 75 mg/m2 on days 1-5
  * Dose level 3: azacitidine 55 mg/m2 on days 1-5
  * Dose level 4: azacitidine 75 mg/m2 on days 1-5
  Each cycle = 28 days. Subjects may receive up to 6 cycles.
  vorinostat: • Dose level 1: oral vorinostat at 300 mg BID on Days 1-7.
  * Dose level 2: oral vorinostat at 200 mg BID on Days 1-7.
  * Dose level 3: oral vorinostat at 300 mg BID on Days 1-14.
  * Dose level 4: oral vorinostat at 200 mg BID on Days 1-14.
  Each cycle = 28 days. Subjects receive up to 6 cycles.
Period: Overall Study
Arm/Group | All Subjects
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 66.5 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR)
Time Frame: 2 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants | 1

ADVERSE EVENTS:
Groups:
- All Subjects: all subjects
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=18)
anemia (Blood and lymphatic system disorders) | 14
thrombocytopenia (Blood and lymphatic system disorders) | 6
leucopenia (Blood and lymphatic system disorders) | 5
neutropenia (Blood and lymphatic system disorders) | 2
nausea (General disorders) | 12
hypoglycemia (Blood and lymphatic system disorders) | 7
renal impairment (Renal and urinary disorders) | 7
diarrhea (Gastrointestinal disorders) | 6
vomiting (General disorders) | 6
raised ALP (Blood and lymphatic system disorders) | 5
hyperglycemia (Blood and lymphatic system disorders) | 5
fatigue (General disorders) | 4
fever (General disorders) | 3
hyperbilirubinemia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes